CLINICAL TRIAL: NCT05779436
Title: Real-Time Cholangioscopy Artificial Intelligence Evaluation of Biliary Strictures
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vinay Chandrasekhara, Principal Investigator, Mayo Clinic
Other Study IDs: 23-000450
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Biliary Stricture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing cholangioscopy for evaluation biliary stricture

SUMMARY:
The purpose of this study is to demonstrate the feasibility and validity of a previously developed peroral cholangioscopy (POC) convolutional neural network (CNN) to determine the etiology of biliary strictures when used in real-time.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Anticipation that patient may undergo POC during an endoscopic retrograde cholangioscopy
* Pregnant patients can be included in the study. Use of the POC-CNN does not convey any new risk to the patient nor fetus.
* Non-English speaking subjects will be included in the study. Consent for the procedure itself is always done with the assistance of an interpreter via telephone or video. Use of the POC-CNN will be discussed with all patients via this interpreter during the procedure consent.

Exclusion Criteria:

* Age <18 years old
* No indication that cholangioscopy will be performed during endoscopic retrograde cholangiopancreatography (ERCP)
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biliary strictures who are undergoing peroral cholangioscopy (POC) during endoscopic retrograde cholangiopancreatography (ERCP) for the evaluation of a biliary strictures will be identified via review of procedure listings at Mayo Clinic Rochester, Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
POC-CNN Model AUC | Patients will be considered negative for malignancy only with 12 months of negative follow-up or definitive negative surgical histology.
  Area Under the Curve (AUC) analysis for POC-CNN for classification of malignant biliary stricture

SECONDARY OUTCOMES:
Test characteristics of POC-CNN | Patients will be considered negative for malignancy only with 12 months of negative follow-up or definitive negative surgical histology.
  Sensitivity and Specificity of POC-CNN for the diagnosis of malignant biliary stricture, Sensitivity and Specificity of biliary brushings and biliary biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Chandrasekhara, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Massachusetts, Worcester, Massachusetts
  - Mayo Clinic Minnesota, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials